CLINICAL TRIAL: NCT01717222
Title: Effect of Intraperitoneal and Intravenous Lignocaine on Pain Relief Following Laparoscopic Cholecystectomy - A Randomized Clinical Trial
Brief Title: Effect of Intraperitoneal and Intravenous Lignocaine on Pain Relief Following Laparoscopic Cholecystectomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Jawaharlal Institute of Postgraduate Medical Education & Research (Other Government)
Responsible Party: Principal Investigator, Dr.D.Ram, Junior Resident, Jawaharlal Institute of Postgraduate Medical Education & Research
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SEC/2011/4/109
Record Dates: First submitted 2012-10-24; First posted 2012-10-30 (Estimated); Last update posted 2012-10-30 (Estimated); Status verified 2012-10

CONDITIONS: Pain, Postoperative; Analgesic Requirement; Stress Response; Return of Bowel Activity; Inadequate or Impaired Respiratory Function
Keywords: Lignocaine; Laparoscopic cholecystectomy; Pain relief
MeSH Terms: conditions — Pain, Postoperative; Fractures, Stress; Respiratory Insufficiency | interventions — Lidocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intraperitoneal (IP) group (Active Comparator): Patients will receive 100 ml of 0.2% Lignocaine as intraperitoneal lignocaine irrigation in the gall bladder fossa along with a placebo of normal saline of volume equivalent to 1.5 mg/kg of intravenous lignocaine at induction and normal saline of volume equivalent to 2 mg/kg/hour of intravenous lignocaine as continuous infusion until one hour postoperatively to ensure blinding
  Interventions: Drug: Intraperitoneal Lignocaine
- Intravenous (IV) group (Active Comparator): Patients will receive 1.5mg/kg of intravenous lignocaine as bolus dose at induction and 2mg/kg/hour as continuous infusion of intravenous lignocaine until one hour after surgery and 100 ml of saline intraperitoneally as placebo to ensure blinding.
  Interventions: Drug: Intravenous Lignocaine

INTERVENTIONS:
Drug: Intraperitoneal Lignocaine — Patients will receive 100 ml of 0.2% lignocaine
  Other Names: IP Lignocaine
  Arms: Intraperitoneal (IP) group
Drug: Intravenous Lignocaine — Intravenous group patients will receive 1.5mg/kg of lignocaine as bolus dose at induction and 2mg/kg/hour as continuous infusion until one hour after surgery
  Other Names: IV lignocaine
  Arms: Intravenous (IV) group

SUMMARY:
Laparoscopic Cholecystectomy is the treatment of choice for patients with symptomatic gall stones. For pain relief following laparoscopic cholecystectomy both intraperitoneal and intravenous administration of lignocaine has been used. But it is not clear from the existing literature which form of administration is more effective for pain relief. Hence this study has been undertaken with the following hypothesis : Intravenous lignocaine is superior to intraperitoneal lignocaine for postoperative pain relief and minimizing the stress response in laparoscopic cholecystectomy.

DETAILED DESCRIPTION:
Laparoscopic Cholecystectomy is the treatment of choice for patients with symptomatic gall stones. For pain relief following laparoscopic cholecystectomy both intraperitoneal and intravenous administration of lignocaine has been used. But it is not clear from the existing literature which form of administration is more effective for pain relief. Hence this study has been undertaken with the following hypothesis : Intravenous lignocaine is superior to intraperitoneal lignocaine for postoperative pain relief and minimizing the stress response in laparoscopic cholecystectomy.

In this study the effect of intraperitoneal and intravenous lignocaine will be assessed based on the postoperative pain scores, total analgesic requirement, stress response in the form of total leukocyte count, c-reactive protein levels,return of bowel activity.

ELIGIBILITY:
Inclusion Criteria:

* Patients planned for elective laparoscopic cholecystectomy in the age group of 20 -60 years belonging to American society of anesthesiologists (ASA)score I-II

Exclusion Criteria:

* Chronic pain diseases other than gall stone disease.
* Use of opioids, steroids, Non steroidal anti inflammatory drugs or alcohol.
* Allergy and contraindication to Lignocaine.
* Conversion to open cholecystectomy.
* Patients who do not comprehend Visual analogue scale (VAS) / patient controlled analgesia (PCA).

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2011-12; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Post operative pain relief | 1 hour postoperatively
  Post operative pain relief will be assessed by visual analogue scale with values between 0 and 10. 0 denotes no pain and 10 denotes worst pain. the patient uses this scale to represent his/her pain at 1 hour postoperatively.

SECONDARY OUTCOMES:
Postoperative Analgesic Requirement | First 24 hours in the postoperative period
  Patients will get analgesia through patient controlled analgesia pump (PCA). This pump delivers Morphine for pain relief. This will be delivered at 1 mg/ml bolus dose with a lock out period of 15 minutes without any background infusion of the drug. The total requirement over a period of 24 hours will be noted. Also the time taken for the patient to take the first analgesic dose will be recorded. The total demands and the number of good demands in the PCA pump will also be recorded.
Postoperative pain relief | 8 hours postoperatively
  Post operative pain relief will be assessed by visual analogue scale with values between 0 and 10. 0 denotes no pain and 10 denotes worst pain. the patient uses this scale to represent his/her pain at 8 hours postoperatively
Postoperative pain relief | 24 hours postoperatively
  Post operative pain relief will be assessed by visual analogue scale with values between 0 and 10. 0 denotes no pain and 10 denotes worst pain. the patient uses this scale to represent his/her pain at 24 hours postoperatively
Postoperative pain relief | 48 hours postoperatively
  Post operative pain relief will be assessed by visual analogue scale with values between 0 and 10. 0 denotes no pain and 10 denotes worst pain. the patient uses this scale to represent his/her pain at 48 hours postoperatively

OTHER OUTCOMES:
Stress response in the form of Total Leucocyte Count (TLC) and C- reactive protein (CRP) | Preoperatively and 48 hours Postoperatively
  Blood will be analyzed for TLC and CRP preoperatively and 48 hours postoperatively to assess the stress response
Respiratory Function | Preoperatively and 48 hours Postoperatively
  Respiratory function will be assessed by measuring the peak expiratory flow rate (PEFR)at the above mentioned time frames.
Return of bowel activity | upto to 48 hours
  This will be assessed by asking the time at which the patient perceives the first bowel movement and also the time for passage of flatus post surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Sarath Chandra Sistla, M.S.,, Study Chair — Jawaharlal Institute of Postgraduate Medical Education & Research
Locations (1):
- Department of Surgery, JIPMER, Puducherry, Puducherry, India

REFERENCES:
- [Background] Jabbour-Khoury SI, Dabbous AS, Gerges FJ, Azar MS, Ayoub CM, Khoury GS. Intraperitoneal and intravenous routes for pain relief in laparoscopic cholecystectomy. JSLS. 2005 Jul-Sep;9(3):316-21. PMID 16121879
- See also: Pubmed site — http://www.ncbi.nlm.nih.gov